CLINICAL TRIAL: NCT02404818
Title: UFPTI 1431 - HL02: Investigating Early Markers of Radiation-Induced Cardiac Injury in Hodgkin Lymphoma Survivors Treated With Either Photon or Proton Radiation
Brief Title: Early Markers of Radiation-Induced Cardiac Injury in Hodgkin Lymphoma Treated With Radiation Therapy
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: UFPTI-1431-HL02; IRB201703302 (Other: UF IRB-03)
Record Dates: First submitted 2015-03-20; First posted 2015-04-01 (Estimated); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Hodgkin's Lymphoma
Keywords: Radiation; Cardiac; Hodgkin's lymphoma
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Survivors of Hodgkin's lymphoma: Cardiac Magnetic Resonance Imaging and Echocardiogram
  Interventions: Procedure: Cardiac Magnetic Resonance Imaging; Procedure: Echocardiogram

INTERVENTIONS:
Procedure: Cardiac Magnetic Resonance Imaging — A cardiac MRI will be performed.
Procedure: Echocardiogram — An echocardiogram will be performed for the following information: M-mode, two-dimensional, Doppler blood flow measurements, and longitudinal strain and strain rate imaging

SUMMARY:
The purpose of this study is to evaluate if radiation and chemotherapy treatment cause cardiac abnormalities among survivors of Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Completed radiation and chemotherapy treatment for Hodgkin lymphoma involving the mediastinum.
* Patient must be ≥ 18 years at time of consent.

Exclusion Criteria:

* Pregnant women at time of Cardiac MRI
* Contraindications to Cardiac MRI (contrast allergy, metal implants, medical devices)
* Glomerular filtration rate (GFR) < 30, unless approved by Radiologist (UF Health Jacksonville Radiology Policy: Administration of Gadolinium-Based Contrast Agents).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hodgkin's lyphoma survivors that have received radiation at UF Health Proton Therapy Institute and also received chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2015-04; Primary Completion 2021-04-14 (Actual); Study Completion 2021-04-14 (Actual)

PRIMARY OUTCOMES:
Cardiac Abnormalities As Measured By Cardiac MRI | Day 1
Cardiac Abnormalities As Measured By Echocardiogram | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Bradford S Hoppe, MD, MPH, Principal Investigator — University of Florida Health Proton Therapy Institute
Locations (1):
- University of Florida Health Proton Therapy Institute, Jacksonville, Florida, United States